CLINICAL TRIAL: NCT04696991
Title: The Effect of Pecha-Kucha Method on the Discharge Readiness and Anxiety Levels: A Randomized Controlled Trial
Brief Title: Effect of the Pecha-Kucha Method on the Discharge Readiness and Anxiety Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysegul Durmaz (Other)
Responsible Party: Sponsor-Investigator, Aysegul Durmaz, Asst. Prof., Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P-K Met. Dis. and Anx.
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Anxiety; Post Procedural Discharge; PechaKucha Method
Keywords: PechaKucha; Postpartum Discharge; Anxiety; Mobile Phone
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The research is a single-blind randomized controlled experimental study. In view of the two groups called E and C, the total number of blocks was calculated as 20 blocks and the number of the participant mothers per block was calculated as 12 mothers, namely, 6 mothers for group E and 6 mothers for group C. Through MS Office Excel 2013, 13 numbers were randomly selected from among numbers from 1 to 20 (9, 17, 19, 4, 14, 3, 14, 1, 20, 16, 12, 8, 20, 2, and 5). By ensuring that each group has 78 mothers, a total of 156 mothers were assigned to experimental and control groups in equal numbers and homogeneously.
  In this context, the research was completed with the participation of 140 mothers, namely, 70 mothers in the experimental group and 70 mothers in the control group.
Who Masked: Participant
Masking Description: Participants didn't know which group they were allocated. The participants will be blind when they take postpartum discharge training with PechaKucha method from investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The mothers in the experimental group (70) were given the postpartum discharge education with PechaKucha Method.
  Interventions: Behavioral: The postpartum discharge education with PechaKucha Method.
- Control Group (No Intervention): The mothers in the control group (70) were given the routine postpartum discharge education.

INTERVENTIONS:
Behavioral: The postpartum discharge education with PechaKucha Method. — The postpartum discharge training in which the PechaKucha method was applied via the smartphones was offered to the mothers in the experimental group whereas the mothers in the control group had solely the routine discharge training. The postpartum training was offered as per the Postpartum Care Management Guideline of the Ministry of Health of Turkey. The discharge training was offered to the experimental group by using the PechaKucha presentation technique.
  Arms: Experimental Group

SUMMARY:
H1a: Between the women receiving discharge training with the PechaKucha method by using smartphones and the women taking the routine discharge training in the early postpartum period, there is a statistically significant difference in the discharge readiness levels.

H1b: Between the women receiving discharge training with the PechaKucha method by using smartphones and the women taking the routine discharge training in the early postpartum period, there is a statistically significant difference in the anxiety levels.

H0a: Between the women receiving discharge training with the PechaKucha method by using smartphones and the women taking the routine discharge training in the early postpartum period, there is no statistically significant difference in the discharge readiness levels.

H0b: Between the women receiving discharge training with the PechaKucha method by using smartphones and the women taking the routine discharge training in the early postpartum period, there is no statistically significant difference in the anxiety levels.

DETAILED DESCRIPTION:
The research was conducted as a single-blind controlled study with simple random sampling. It was carried out at a tertiary-level hospital in Turkey in February-August 2019.

The research population was composed of the mothers who had cesarean delivery at the maternity service of a tertiary-level hospital in Turkey. The size of the research sample was calculated with power analysis. Considering the likelihood that some participants would later be excluded from the research or leave it, a total of 156 mothers who met the inclusion criteria for the research were assigned to the experimental group (78) and control group (78).

Both the experimental and control groups each had 78 mothers, and hence, a total of 156 mothers were included in the study. The postpartum discharge training in which the PechaKucha method was applied via the smartphones was offered to the mothers in the experimental group whereas the mothers in the control group had solely the routine discharge training. The research was completed with the participation of 140 mothers, namely, 70 mothers in the experimental group and 70 mothers in the control group. The discharge training which was comprised of 20 slides created as per the PechaKucha method was offered to the mothers in the experimental group via smartphones. Each slide was displayed for 20 seconds. The presentation took 6 minutes 40 seconds in total. The Q&A session was performed after the presentation. While care was provided and the follow-up activities were performed in the process following the discharge training, feedback about the discharge training topics was received from both groups, discharge training topics were reminded to both groups and the questions of the mothers in both groups were answered.

The 'Personal Information Form', the 'Readiness for Hospital Discharge Scale - New Mother Form', and the 'State-Trait Anxiety Inventory' were used for gathering the research data.

In the statistical analysis, the SPSS (Statistical Package for Social Science) 22.0 software was utilized. Descriptive statistics (mean, standard deviation, frequency, percentage) were used in the evaluation of the findings. Kolmogorov-Smirnov test was employed for identifying whether the research data were normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* To receive postpartum discharge training with PechaKucha method
* To have cesarean birth
* To have singleton birth
* To be within the early postpartum period (the first 48 hours)
* Not have complications at childbirth
* Not have chronic diseases or mental disorders
* Older than 18 years
* To voluntary to participate
* To know how to read, write and speak in Turkish
* To stay within this study until the end
* To fully complete questionnaire
* To have a newborn with no complications
* To have a healthy baby

Exclusion Criteria:

* To receive routine postpartum discharge training
* Not have cesarean birth
* Having multiple birth
* Not to be within the early postpartum period (the first 48 hours)
* Having complications at childbirth
* Having chronic diseases or mental disorders
* Younger than 18 years
* To refuse to participate
* Not knowing how to read, write and speak Turkish
* To leave early this study
* Not fill the questionnaire
* Having a newborn with complications
* Having a baby in need of medical care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Pre-Test Readiness for Postpartum Discharge | the pretest was applied in the first 8-12 hours in the postpartum period.
  Perceived Readiness for Discharge After Birth Scale-Form for New Mothers (PRDABS-FNM); This is a scale assessing the readiness for discharge by mothers' perceptions. It consists of four subdimensions and 23 items. The first item is answered dichotomously (yes/no). The items between 2 and 23 are calculated through the Likert type points ranging from 0 to 10. The subdimensions consisted of 1. Care skills, 2. Expected support; 3. Strength and ability to cope; 4. Stress control and knowledge of accessing help. The lowest and highest scores are 0 and 220. High scores indicate women's readiness for discharge.
Pre-Test Anxiety Level | the pretest was applied in the first 8-12 hours in the postpartum period.
  State-Trait Anxiety Inventory (STAI): The scale which was developed in 1970 by Spielberger, Gorsuch, and Lushene is comprised of two parts for measuring state anxiety and trait anxiety. Each part has 20 items. The STAI-State is scored as per the severity level of the emotions and behaviors (1: Not at all, 2: Somewhat, 3: Moderately so, and 4: Very much so). In the STAI-State, there are ten reverse-scored items (Items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20). The items of the STAI-Trait are scored as per the expression frequency of the emotions and behaviors (1: Almost never, 2: Sometimes, 3: Often, and 4: Almost always). In the STAI-Trait, there are seven reverse-scored items (Items 21, 26, 27, 30, 33, 36, and 39). In the scoring, two separate keys are prepared for identifying the total weighted values of the straight-scored and reverse-scored items. These constant values are 50 and 35 respectively for the STAI-State and STAI-Trait.

SECONDARY OUTCOMES:
Post-Test Readiness for Postpartum Discharge | the post-test was applied in the first 36-40 hours in the postpartum period.
  Perceived Readiness for Discharge After Birth Scale-Form for New Mothers (PRDABS-FNM); This is a scale assessing the readiness for discharge by mothers' perceptions. It consists of four subdimensions and 23 items. The first item is answered dichotomously (yes/no). The items between 2 and 23 are calculated through the Likert type points ranging from 0 to 10. The subdimensions consisted of 1. Care skills, 2. Expected support; 3. Strength and ability to cope; 4. Stress control and knowledge of accessing help. The lowest and highest scores are 0 and 220. High scores indicate women's readiness for discharge.
Post-Test Anxiety Level | the post-test was applied in the first 36-40 hours in the postpartum period.
  State-Trait Anxiety Inventory (STAI): The scale which was developed in 1970 by Spielberger, Gorsuch, and Lushene is comprised of two parts for measuring state anxiety and trait anxiety. Each part has 20 items. The STAI-State is scored as per the severity level of the emotions and behaviors (1: Not at all, 2: Somewhat, 3: Moderately so, and 4: Very much so). In the STAI-State, there are ten reverse-scored items (Items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20). The items of the STAI-Trait are scored as per the expression frequency of the emotions and behaviors (1: Almost never, 2: Sometimes, 3: Often, and 4: Almost always). In the STAI-Trait, there are seven reverse-scored items (Items 21, 26, 27, 30, 33, 36, and 39). In the scoring, two separate keys are prepared for identifying the total weighted values of the straight-scored and reverse-scored items. These constant values are 50 and 35 respectively for the STAI-State and STAI-Trait.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: If study' IPD are used, my article should be cited.

REFERENCES:
- [Background] McCarter-Spaulding D, Shea S. Effectiveness of Discharge Education on Postpartum Depression. MCN Am J Matern Child Nurs. 2016 May-Jun;41(3):168-72. doi: 10.1097/NMC.0000000000000236. PMID 27128643
- [Background] Yonemoto N, Dowswell T, Nagai S, Mori R. Schedules for home visits in the early postpartum period. Cochrane Database Syst Rev. 2017 Aug 2;8(8):CD009326. doi: 10.1002/14651858.CD009326.pub3. PMID 28770973
- [Background] Tiruneh GT, Shiferaw CB, Worku A. Effectiveness and cost-effectiveness of home-based postpartum care on neonatal mortality and exclusive breastfeeding practice in low-and-middle-income countries: a systematic review and meta-analysis. BMC Pregnancy Childbirth. 2019 Dec 18;19(1):507. doi: 10.1186/s12884-019-2651-6. PMID 31852432
- [Background] Ramos-Rincon JM, Sempere-Selva TS, Romero-Nieto M, Peris-Garcia J, Martinez-de la Torre G, Harris M, Fernandez-Sanchez J. Pecha Kucha presentations by medical students in Spain. Int J Med Educ. 2018 Sep 19;9:244-245. doi: 10.5116/ijme.5b92.52e3. No abstract available. PMID 30244236
- [Background] Saracoglu KT, Yilmaz M, Turan AZ, Kus A, Colak T, Saracoglu A. Pecha Kucha with Part-Task Training Improves Airway Management in Fresh Frozen Cadavers: A Case-Control Observational Study. Med Princ Pract. 2020;29(6):532-537. doi: 10.1159/000506597. Epub 2020 Feb 19. PMID 32069469
- [Background] Ramos-Gallardo G, Mecott-Rivera GA, Limon-Cervantes R, Garcia-Perez M, Rodriguez-Olivares E. How to Improve Speaking Skills in Plastic Surgery Training? Survey in Residents Participants in Pecha Kucha Contest. World J Plast Surg. 2018 May;7(2):166-170. PMID 30083498
- [Background] Pawluski JL, Lonstein JS, Fleming AS. The Neurobiology of Postpartum Anxiety and Depression. Trends Neurosci. 2017 Feb;40(2):106-120. doi: 10.1016/j.tins.2016.11.009. Epub 2017 Jan 24. PMID 28129895
- [Background] Nakic Rados S, Tadinac M, Herman R. Anxiety During Pregnancy and Postpartum: Course, Predictors and Comorbidity with Postpartum Depression. Acta Clin Croat. 2018 Mar;57(1):39-51. doi: 10.20471/acc.2017.56.04.05. PMID 30256010
- [Derived] Gun Kakasci C, Durmaz A. A creative and practical approach to postpartum discharge education: Pecha Kucha training via smart phone. Health Care Women Int. 2022 Dec;43(12):1482-1502. doi: 10.1080/07399332.2022.2043860. Epub 2022 Jun 21. PMID 35726861